CLINICAL TRIAL: NCT06068231
Title: A Prospective Clinical Study to Evaluate the Outcome of Early Loading of Implants in the Maxillary Anterior Region With Alveolar Bone Defects
Brief Title: A Study of Early Loading of Implants in the Maxillary Anterior Region With Alveolar Bone Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Entang Wang, Attending, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHZhejiangU#2022(073)
Record Dates: First submitted 2023-08-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Dental Implant
Keywords: Alveolar Bone Defects; Early Loading of Dental Impalnt; Dental Impalnt treatment
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study takes a single-blind method. During research process, the researchers and paticipant cannot avoid knowing the time of loading during the clinical examination and operation, so the outcomes assessor can only be single-blinded.The clinical examination data were measured and averaged by two independent clinicians. The data was analysed by a third person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early loading group (Experimental): Early Loading Group: Implants were loaded with temporary restorations between 48 hours and 3 months after implantation and had occlusal contact with opposing dentition. The early loading time point was set at 6-8 weeks after implantation in this study.
  Interventions: Device: Temporary Crown
- Conventional Loading Group (Active Comparator): Implants were loaded at least 3 months after implantation and had occlusal contact with opposing dentition.
  Interventions: Device: Permanent Crown

INTERVENTIONS:
Device: Temporary Crown — Implants were loaded with temporary restorations 6 to 8 weeks after implantation and had occlusal contact with opposing dentition.
  Other Names: Early Loading
  Arms: early loading group
Device: Permanent Crown — Implants were loaded with permanent restorations at least 3 months after implantation and had occlusal contact with opposing dentition.
  Other Names: Conventional Loading
  Arms: Conventional Loading Group

SUMMARY:
With the improvement of people's living standards, implant restoration has become an ideal method for partially and completely edentulous patients. Traditional classic implant theory suggests a 3-6 month undisturbed healing period is required before permanent loading can take place. However, this loading plan takes a long time and cannot timely meet the chewing function and aesthetic needs of patients with anterior maxillary tooth loss. Currently, with the continuous improvement of implant design and surface treatment techniques, the speed of implant-bone integration has been increasing, and early loading has gradually become a clinical option.

After carefully reviewing the research conducted by domestic and international scholars on early loading of implants in the anterior maxillary region , we found that the cases included in the articles were patients with anterior maxillary tooth loss who did not require simultaneous guided bone regeneration (GBR) surgery. It is well known that patients with anterior maxillary tooth loss often have significant alveolar bone defects. In such cases, GBR techniques are commonly used to repair the bone defect. However, due to the lack of relevant studies, the clinical loading strategies for implant cases with accompanying bone defects are relatively conservative. Clinically, a delayed loading restoration strategy is usually employed, which typically requires a delay of 6 months or even longer.

However, delayed loading increases the patient's edentulous time, affects the function and stability of the dental arch, and increases the patient's psychological burden. Therefore, whether an early loading strategy can be used for implant cases with alveolar bone defects in the anterior maxillary region has become a key issue in clinical practice. However, there is few research reported on the timing and effectiveness of early loading of implants in the anterior maxillary region with accompanying alveolar bone defects.

This study aims to evaluate the clinical effects of early loading in patients with anterior maxillary single-wall bone defects through a prospective clinical randomized controlled trial.

DETAILED DESCRIPTION:
1. Research Objectives

   This study aims to compare the marginal bone resorption, implant success rate, complication rate, soft tissue condition, and patient satisfaction between early loading and conventional loading of implants in the maxillary anterior region with alveolar bone defects using a combination of prospective clinical control study and three-dimensional finite element analysis. The study aims to explore the clinical effects of early loading of implants in the maxillary anterior region with alveolar bone defects and provide clinical evidence for early loading of implants in this area.
2. Research Design and Methods

2.1 Subject Inclusion Criteria, Exclusion Criteria, and Grouping Criteria According to the purpose of the study, prospective intervention single-center randomized clinical trial was designed. Patients treated with implant restoration in the Oral Implant Center of Stomatology Hospital Affiliated to Zhejiang University School of Medicine, from July 2022 to June 2025 were recruited. The recruited patients were divided into the early loading group with bone defects (referred to as the early loading group) and the conventional loading group with bone defects (referred to as the conventional loading group).

2.1.1Inclusion Criteria: (1)Age: 18-60 years; (2)Gender: Male or Female; (3)Patients with a single missing upper anterior tooth and a labial open-type single-wall bone defect who underwent simultaneous guided bone regeneration (GBR) surgery; (4)Patients choosing the ITI implant system; (5)Patients without a history of systemic diseases such as cardiovascular disease, hypertension, diabetes, etc.;(6)Patients with no history of periodontal disease or have undergone periodontal treatment and can maintain good oral hygiene with no smoking history; (7)Patients without a history of radiation therapy, hepatitis, tuberculosis, or any familial hereditary diseases; (8)Patients with a normal anterior occlusion

Exclusion Criteria:

(1) Patients with bone defects other than labial open-type single-wall bone defects in the anterior region; (2) Patients with multiple consecutive missing upper anterior teeth; (3) Patients with a history of systemic diseases, infectious diseases, or familial hereditary diseases;(4) Patients with poor oral hygiene; (5) Patients with bruxism or teeth clenching.

2.1.2 Grouping Criteria

Early Loading Group: Implants were loaded with temporary restorations between 48 hours and 3 months after implantation and had occlusal contact with opposing dentition. The early loading time point was set at 6-8 weeks after implantation.

Conventional Loading Group: Implants were loaded at least 3 months after implantation and had occlusal contact with opposing dentition.

2.2 Subject Withdrawal Criteria and Trial Termination Criteria: During the trial, participants had the right to withdraw at any stage without affecting their relationship with the doctors or access to medical services. If a participant was terminated from the trial, it would not affect their routine treatment. The anticipated reasons for trial termination include: (1）Participants not following the doctor's instructions (2）Participants experiencing serious conditions requiring treatment (3）The research doctor deems that terminating the study is in the best interest of the participant's health and well-being.

2.3 Clinical Procedures

2.3.1 Surgical Procedure: After undergoing routine disinfection, the subjects received local anesthesia. The implant was placed in the optimal position, with bone grafting at the labial single-wall bone defect. A membrane was then applied and tension-free suturing was utilized. Relevant information such as tooth position, single-wall bone defect height and width, and implant dimensions were recorded. Implant stability quotient (ISQ) and torque values were measured, and antibiotics were administered for three days.

2.3.2 Restorative Procedure: Postoperative follow-up visits were scheduled regularly. ISQ values of the implants were measured and recorded. At 6-8 weeks after implantation, if the measured ISQ value was ≥65, the early loading group received temporary restorations. If the measured ISQ value was <65, weekly follow-up visits were continued until the ISQ value reached ≥65 for the conventional loading group. Permanent restorations were performed for the early loading group at 3-4 months after implantation.

2.4 . Design plan and expected duration and specific arrangements for participating in clinical trials: Subjects are expected to participate in clinical trials for 2 years, and need to complete follow-up. Measure the ISQ value and torque value of the implant on the day of surgery. ISQ value is also measured on the six weeks after surgery, 3months, 6 months and 1year after loading .Examine the condition of the implant restoration and soft tissues on the 3months, 6 months and 1year after loading .Evaluate patient satisfaction at 1 year after loading . Imaging examinations, including parallel projection X-rays and CBCT, are required on the day of surgery, 3months, 6 months, and 1-2years after loading.

2.5 Main and Secondary Outcome Measures

The main outcome measure of this study is the marginal bone resorption around the implants. The secondary outcome measures include implant success rate, complication rate, PES index, gingival index, bleeding on probing, pocket probing depth, and patient satisfaction.

3.Sample Size Calculation

This study adopts a non-inferiority test, with a 1:1 ratio of samples between the experimental group and the control group. The critical value is defined as 0.5mm, indicating that the experimental group's marginal bone resorption should not exceed 0.5mm compared to the control group. The reference literature reported a marginal bone resorption of 1.0±0.6mm in the control group after 18 months of conventional loading.

Using the formula:

n=((Z_(1-α)+Z_(1-β) )^2×(σ_1^2+σ_2^2 ))/(ε-δ)^2

With the application of PASS2021 software, a minimum of 32 cases were required. Considering a dropout rate of 20%, the sample size was set at 40 cases per group.

4. Data Management and Confidentiality

Each subject enrolled in the study will be assigned a unique number, with the experimental group numbered as (T1, T2, T3, etc.) and the control group numbered as (C1, C2, C3, etc.). The data record forms do not contain personal privacy information of the subjects. Only research personnel, ethics committee, and relevant management departments have access to the data. If a subject withdraws or is terminated from the trial, the related data and information will be discarded. Records of subject identities will be kept confidential, and these data will not be disclosed outside of the relevant legal and/or regulatory requirements. Experimental data will be managed using Excel 2013 for data collection through clinical case data compilation and calculation, inquiry, and questionnaire surveys, with regular backups. For missing data, mean values, weighted means, medians, etc., will be used to fill in numerical data. For categorical data, the most common values will be used for completion. Unused and illogical data will be discarded. The data of the subjects used for statistical analysis should be complete and accurate.

5.Informed Consent

This study does not involve vulnerable populations. All subjects will sign an informed consent form. The specific process is as follows: When patients first visit the Implant Department ,the researchers will provide information and obtain informed consent from the subjects. (1) Based on the subjects' cultural level, the research doctors will explain the research background, purpose, significance, steps, potential benefits and risks, research duration, requirements for cooperation, cost coverage, compensation and treatment in case of harm during the trial, and confidentiality regulations. (2) After the subjects have a preliminary understanding of the trial information and basic agreement, they will be provided with an easy-to-understand informed consent form that has been approved by the ethics committee. The verbal information will be supplemented in the written informed consent form. The subjects will be asked to read the informed consent form and given sufficient time to read and inquire about the details of the study and any other questions they may have, in order to make an independent decision on whether or not to participate in the study. (3) If a subject lacks the capacity or is unable to give informed consent fully, they will not be recruited as subjects. (4)Throughout the process, the principles of voluntariness will be upheld, the subjects' privacy will be respected, no deception, excessive persuasion, or coercion will be used, and detailed answers will be provided to the subjects and their families, giving them sufficient time to fully understand the entire study. Whether or not to participate is entirely up to the subjects' own will. After signing the informed consent form, the subjects will formally join the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years;
2. Gender: Male or Female;
3. Patients with a single missing upper anterior tooth and a labial open-type single-wall bone defect who underwent simultaneous guided bone regeneration (GBR) surgery;
4. Patients choosing the ITI implant system;
5. Patients without a history of systemic diseases such as cardiovascular disease, hypertension, diabetes, etc.;
6. Patients with no history of periodontal disease or have undergone periodontal treatment and can maintain good oral hygiene with no smoking history;
7. Patients without a history of radiation therapy, hepatitis, tuberculosis, or any familial hereditary diseases;
8. Patients with a normal anterior occlusion.

Exclusion Criteria:

1. Patients with bone defects other than labial open-type single-wall bone defects in the anterior region;
2. Patients with multiple consecutive missing upper anterior teeth;
3. Patients with a history of systemic diseases, infectious diseases, or familial hereditary diseases;
4. Patients with poor oral hygiene;
5. Patients with bruxism or teeth clenching.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
marginal bone resorption | 1-2years
  The degree of bone resorption at the shoulder edge of the implant. Bone level was measured by a single reader on CBCT taken after implant surgery, temporary restoration, final restoration, and at the 12-month follow-up.

SECONDARY OUTCOMES:
Implant Success Rate | 1-2years
  Implant success were assessed at suture removal, provisional restoration, final restoration, and at the 12-month follow-up. Implant success was defined according the criteria by Buser et al. ,i.e., absence of pain, foreign body discomfort or dysesthesia, absence of recurrent peri-implant infection with suppuration, absence of implant mobility, and absence of continuous peri-implant radiolucency.
Complication rate | 1-2years
  Complication were assessed at suture removal, provisional restoration, final restoration, and at the 12-month follow-up. Complication was defined Implant fracture，loose crowns and crowns breakage.
PES index | 1-2years
  peri-implant soft tissue index (PES). the PES comprises the following five variables : mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue color and texture at the facial aspect of the implant site. A score of 2, 1, or 0 is assigned to all five PES parameters. The five described parameters (5×2) add up, under optimum conditions, to a score of 10; the threshold of clinical acceptability was set at 6.
probing depth | 1-2years
  periodontal examination, in the form of probing depth (PD) , was performed at pre-screening ,final restoration and at the 12-month follow-up.
probing bleeding index | 1-2years
  periodontal examination, in the form of bleeding on probing (BoP), was performed at pre-screening ,final restoration and at the 12-month follow-up.
Satisfaction assessed by the VAS | 1-2years
  Patients answered five questions regarding their satisfaction on five parameters: prosthesis comfort, aesthetics, ability to chew, pronunciation and stability. Patients were asked to mark for each question the respective Visual Analog Scale (VAS) which is a 100 mm straight horizontal line with the left end indicating "not at all satisfied" and the right end "very satisfied". The satisfaction value was determined by the distance from the left end of the scale to the mark in millimeters and expressed as percentage (10 mm corresponds to 10%, 20 mm 20%, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Yixun Chen, Principal Investigator — Stomatology Hospital Affiliated to Zhejiang University School of Medicine
Locations (1):
- Stomatology Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No